CLINICAL TRIAL: NCT02365870
Title: Anxiety in Parkinson's: Use of Quantitative Methods to Guide Rational Treatment
Acronym: ANXPD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding cycle completed
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00092051; 1K23AG044441-01A1 (NIH)
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Anxiety Disorders; Parkinson Disease
Keywords: Anxiety Disorders; Parkinson Disease; rotigotine
MeSH Terms: conditions — Anxiety Disorders; Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rotigotine (Active Comparator): rotigotine transdermal patch 2mg to 6mg daily per 24 hour patch for 8 weeks
  Interventions: Drug: rotigotine transdermal patch
- placebo (Placebo Comparator): placebo transdermal patch 2mg to 6mg daily per 24 hour patch for 8 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rotigotine transdermal patch — Participants will receive the dopamine agonist rotigotine in the form of a transdermal patch to be worn daily
  Other Names: Neupro
  Arms: rotigotine
Drug: placebo — Participants will receive a placebo transdermal patch to be worn daily
  Other Names: placebo control
  Arms: placebo

SUMMARY:
This study will evaluate the effectiveness of the rotigotine transdermal patch in reducing anxiety in people with Parkinson's disease.

DETAILED DESCRIPTION:
Anxiety is a serious medical condition that worsens quality of life by negatively affecting peoples thoughts, feelings, and ability to function normally. Anxiety can affect anyone, but people with Parkinson's appear to be at a much higher risk with an estimated 40% or more suffering from anxiety. Parkinson's is a neurological disorder that causes tremor and other problems with normal movements. The disease symptoms are believed to be caused in large part by the loss of dopamine producing cells in the midbrain. Anxiety in Parkinson's may be associated with the loss of dopamine caused by the disease and therefore may respond to dopamine based treatments. This study will evaluate the effectiveness of the rotigotine transdermal patch, a dopamine replacement medication, in reducing symptoms of anxiety in people with Parkinson's disease.

Participants in this double-blind study will be randomly assigned to receive either rotigotine or a placebo patch for 8-weeks. All participants will be evaluated at the study site at baseline and weeks 2, 4, and 8. Psychiatric, cognitive, and movement assessments will be performed along with a review of anxiety symptoms. All participants will be offered continued routine psychiatric care with the study physician upon completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 Anxiety Disorder
* Stable medical history and general health
* On stable anti-parkinsonian therapy for 2 weeks before enrollment

Exclusion Criteria:

* Unstable medical disease of comorbid psychiatric disease
* Dementia
* Subjects with less than one year duration of Parkinson's
* Current treatment with a dopamine agonist

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Pontone, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rotigotine | Placebo
Started | 1 | 3
Completed | 1 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotigotine | Placebo | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (0) | 68.3 (6.4) | 62.75 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Participants with Depression at baseline [Count of Participants; unit: Participants] — The measure reports participants who were found to have depression (score > 7) at baseline per The Hamilton Depression Rating Scale (HAMD). The HAMD is a 17-item questionnaire, with each item assigned a score ranging from 0 ("not present") to 4 ("severe"). The total score of this scale ranges from 0 to 68, with scores greater than 7 indicating mild depressive symptoms.
  Participants | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Anxiety Symptom Severity as Assessed by the Hamilton Anxiety Rating Scale
Description: The main outcome measure for this study was change in anxiety symptom severity over the course of the study. Anxiety severity was measured using the Hamilton Anxiety Rating Scale (HARS).The HARS is a 14-item questionnaire, with each item assigned a score ranging from 0 ("not present") to 4 ("severe"). The total score of this scale ranges from 0 to 56, with scores greater than 17 indicating mild severity, scores between 18 and 24 indicating mild to moderate severity and scores greater than 25 indicating moderate to severe severity.
Time Frame: Baseline, weeks 2, 4 and 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 1 | 3
score on a scale
  Baseline | 23 (0) | 20.7 (5.1)
  Week 2 | 20 (0) | 13.7 (6.4)
  Week 4 | 5 (0) | 18.3 (13.6)
  Week 8 | 9 (0) | 14.7 (11.9)

2. Secondary Outcome: Change in Depression Symptom Severity as Assessed by the 17-item Hamilton Depression Rating Scale
Description: The main outcome measure for this study was change in depression symptom severity over the course of the study. Depression severity was measured using the Hamilton Depression Rating Scale (HAMD). The HAMD is a 17-item questionnaire, with each item assigned a score ranging from 0 ("not present") to 4 ("severe"). The total score of this scale ranges from 0 to 68, with scores greater than 7 indicating mild depressive symptoms.
Time Frame: Baseline, weeks 2, 4 and 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 1 | 3
score on a scale
  Baseline | 10 (0) | 8 (2)
  Week 2 | 10 (0) | 5.3 (1.5)
  Week 4 | 4 (0) | 7.3 (7.1)
  Week 8 | 5 (0) | 4.3 (5.1)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the course of the study. This spanned from baseline through the tapering period for the drug (up to 42 days after the final study visit).
Arm/Group | Rotigotine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=1) | Placebo (N=3)
Excessive Somnolence (General disorders) | 0 (0) | 1 (1) — Mild severity recovered without treatment
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1) — mild severity, not distressing
Edema (Cardiac disorders) | 0 (0) | 1 (1) — mild severity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT02365870/Prot_SAP_000.pdf